CLINICAL TRIAL: NCT03099317
Title: Sinew Acupuncture for Knee Osteoarthritis (KOA): A Randomized, Sham Controlled, Patient and Assessor Blinded, Pilot Trial
Brief Title: Sinew Acupuncture for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UHongKong-UW16-2007
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Sinew Acupuncture; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Intervention Model Description: A randomized sham controlled, single blinded trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be randomized into sinew acupuncture group and sham acupuncture group in a 1:1 ratio.
  Assessors will perform the assessment but not be involved in acupuncture treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sinew acupuncture (Experimental): Subject in the arm will receive real acupuncture intervention.
  Interventions: Other: Sinew acupuncture
- Sham acupuncture (Sham Comparator): Subject in the arm will receive sham acupuncture intervention.
  Interventions: Other: Sham acupuncture

INTERVENTIONS:
Other: Sinew acupuncture — Sinew acupuncture: subject will sit on chair with knee joint flexion with a most comfortable angle nearest to 90 degrees. Acupoints (1-2cm away from the point of tenderness or pain) near the knee will be punctured through the skin by using sterile needles of size 0.30mm × 40mm at the angle of 0-10 degrees pointing along the pain direction and meridian sinew. Immediately, needles will be retreated back just under the skin and inserted 10mm-20mm forward smoothly with minimal pain sensation. Walking and stepping will be advised and governed during acupuncture. The acupoint will be covered with non-allergic bandages to ensure sufficient blinding to the subject. The treatment will last 20 minutes for each session.
  Arms: Sinew acupuncture
Other: Sham acupuncture — Sham acupuncture: subject will receive the same procedures as the sinew acupuncture without penetrating the skin. The needle will be used to puncture on the acupoint slightly without passing through the skin. The acupoint will be covered with non-allergic bandages to ensure sufficient blinding to the subject.
  Arms: Sham acupuncture

SUMMARY:
The study aims to exam whether sinew acupuncture can relieve pain and symptoms of KOA and improve functional movement by Visual Analog Scale (VAS), Western Ontario and McMasters University Osteoarthritis Index (WOMAC), Timed up & Go Test (TUG) and 8-step Stair Climb Test (SCT) assessment, and Quality of life by Short Form-36 (SF-36). A randomized, sham acupuncture controlled, patient and assessor blinded, pilot study will be employed.

DETAILED DESCRIPTION:
Objective:

The proposal aims to examine the efficacy and safety of sinew acupuncture for knee osteoarthritis (KOA).

Hypothesis to be tested:

Sinew acupuncture can reduce pain intensity, and improve knee function and health-related quality of life without significant side effects for KOA subjects compared to a sham acupuncture.

Design:

A randomized, subject- and assessor-blind, sham acupuncture-controlled clinical trial

Participants:

Subjects (N=86) will be randomized into sinew acupuncture or sham acupuncture group (in 1:1 ratio).

Study instrument:

Visual Analog Scale (VAS), Western Ontario and McMasters University Osteoarthritis Index (WOMAC), Timed up & Go Test (TUG), 8-step Stair Climb Test (SCT) assessment, and the Short Form-36 (SF-36).

Intervention:

Sinew acupuncture group will receive 10 sessions of needling in 4 weeks. Sham group will receive the non-invasive intervention with the same procedures. All subjects are followed up for 6 weeks.

Main outcome measures:

VAS for knee pain intensity at week 4 serves as the primary outcome. VAS at other time points, WOMAC score, TUG, SCT and SF-36 will be analyzed as the secondary outcomes.

Data analysis:

Analysis will be on the 'intention to treat' principle. T-test and mixed-effect model analysis will be used to measure primary and secondary outcomes respectively.

Expected results:

Sinew acupuncture treatment can significantly reduce knee pain intensity, and improve knee function and quality of life without obvious side effects.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong permanent residents aged on or above 50, both male and female;
* meet the Clinical Classification Criteria for Osteoarthritis of the Knee by history, physical examination and radiographic findings (recommended by the American College of Rheumatology): history and physical examination: pain in the knee and one of the following (1. Over 50 years of age; 2. Less than 30 minutes of morning stiffness; 3. Crepitus on active motion and osteophytes) and radio graphical findings (Kellgren and Lawrence Grades 2-4):
* with unilateral knee pain or bilateral knee pain;
* in chronic stage (pain of at least 6 month's duration);
* with rated knee pain >40 mm on a visual analog scale (VAS; 0 to 100 mm) within 7 days;
* with X-ray or other radiographic reports are preferable (not necessary);
* who volunteer to participate and sign the consent form;
* able to write and read Chinese.

Exclusion Criteria:

* Patients who are unable to walk;
* with serious infection of knee;
* with suspected tears of ligaments, menisci or acute inflammation of synovial capsule;
* with trauma, ligament damage, fracture, or surgery on the knee(s) within 6 months, as the cause of pain or functional problems (history of knee replacement will be excluded);
* with history of local tumor/malignancy at knee;
* with physical or laboratory findings indicating infection, presence of autoimmune disease or inflammatory arthritis;
* with knee pain caused by radiculopathy / herniation of intervertebral disc;
* with end-stage of diseases and other suspected severe conditions such as deep vein thrombosis of the lower limb, edema related to cancer or cancer treatment, severe blood coagulation disorders, uncontrolled systemic arterial hypertension and severe diabetes;
* with history of prolotherapy, with injections of hyaluronic acid or cortisone within 3 months;
* received acupuncture, electro-acupuncture, Tui-na therapy, massage, physiotherapy for 8 weeks prior to the trial;
* with more severe pain in other regions;
* have severe mental disorders;
* oversensitive to needles;
* insensitive to pain due to advanced diabetes, neuropathy or using strong painkillers;
* fail to be complaint with the treatment protocol.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity measured by VAS | Week 4
  Pain intensity will be measured by VAS

SECONDARY OUTCOMES:
WOMAC | Weeks 0, 1, 2, 3, 4, 6 and 10
  Western Ontario and McMasters University Osteoarthritis Index
TUG | Weeks 0, 2, 4, 6 and 10
  Timed up and go test
8-step SCT | Weeks 0, 2, 4, 6 and 10
  Stair Climb Test
Quality of life measured by SF-36 | Weeks 0, 4, and 10
  Short Form-36

CONTACTS AND LOCATIONS:
Overall Officials: Haiyong Chen, PhD, Principal Investigator — The University of Hong Kong; Kwok Yin Au, PhD, Principal Investigator — The Hong Kong Tuberculosis Association Chinese Medicine Clinic cum Training Centre of the University of Hong Kong
Locations (1):
- The Hong Kong Tuberculosis, Association The University of Hong Kong Clinical Centre for Teaching and Research in Chinese Medicine (Wan Chai), Wan Chai, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lam WC, Au KY, Qin Z, Wu FM, Chong CO, Jiang F, He Y, Ng BFL, Yeung WF, Lao L, Chen H. Superficial Needling Acupuncture vs Sham Acupuncture for Knee Osteoarthritis: A Randomized Controlled Trial. Am J Med. 2021 Oct;134(10):1286-1294.e2. doi: 10.1016/j.amjmed.2021.05.002. Epub 2021 Jun 11. PMID 34126097
- [Derived] Au KY, Chen H, Lam WC, Chong CO, Lau A, Vardhanabhuti V, Mak KC, Jiang F, Lam WY, Wu FM, Chan HN, Ng YW, Ng BF, Ziea ET, Lao L. Sinew acupuncture for knee osteoarthritis: study protocol for a randomized sham-controlled trial. BMC Complement Altern Med. 2018 Apr 23;18(1):133. doi: 10.1186/s12906-018-2195-8. PMID 29685141